CLINICAL TRIAL: NCT03977935
Title: Second-generation Versus First-generation Magnetically Controlled Capsule Gastroscopy for Upper Gastrointestinal Tract: a Randomized Controlled Clinical Trial.
Brief Title: The Second-Generation MCCG for Upper Gastrointestinal Tract.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Clinical Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SG-MCCG-UGT
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2019-06

CONDITIONS: Capsule Endoscopy
Keywords: SG-MCCG; Z-line visualization; Image quality; Gastric examination time; Manipulation performance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The first-generation MCCG group (No Intervention): The patients swallowed the first-generation MCCG with a small amount of water in the left lateral decubitus position. Once the capsule reached the stomach after investigating the esophagus, it was lifted away from the posterior wall, rotated and advanced to the fundus and cardiac regions, and then to the gastric body, angulus, antrum and pylorus. After finishing the stomach examination twice, the endoscopist controlled the capsule to face the pylorus and drag it close to the pylorus. The capsule would enter the duodenal bulb and was held stationary to investigate the duodenal bulb using the "360-degree automatic scanning" mode. In the descending part of duodenum, the endoscopist tried to control the capsule to view the major papilla. After passing through the duodenum, the capsule started to complete the small-bowel examination with the "small-bowel mode". The magnetic steering time for passing through the pylorus was not allowed more than 15 min.
- The second-generation MCCG group (Experimental): All process in this study were the same except that the second-generation capsule (Ankon Navicam-2) was used in the experimental group.
  Interventions: Device: the second-generation MCCG

INTERVENTIONS:
Device: the second-generation MCCG — Patients in the experimental group swallowed the second-generation MCCG (Ankon Navicam-2).
  Arms: The second-generation MCCG group

SUMMARY:
The aim of this study is to evaluate the clinical application of the second-generation MCCG with higher image resolution and frame rate for upper gastrointestinal tract compared with the first-generation.

DETAILED DESCRIPTION:
Magnetically controlled capsule gastroscopy (MCCG) has been widely used in clinical practice for gastric examination. However, there still exist blind spots under MCCG, particularly in the esophagus and duodenum. Although the anatomy of the esophagus and duodenum can be the main cause, MCCG still needs technical improvement. In addition, the gastric examination time under MCCG can be further optimized.

Therefore, a new-generation MCCG is developed with a higher frame rate improved from 0.5-2 to 0.5-8 frames per second, image resolution improved from 480 x 480 to 720 x 720, view angle improved from 140° to 150°, wireless anti-jamming technology is applied as a more effective and stable information transmission method.

This is a prospective, single-centered, blinded randomized controlled pilot study. Subjects receiving MCCG at Changhai Hospital will be randomly allocated into two groups with a ratio of 1:1 before the procedure, the first-generation or the second-generation MCCG. After passage through the esophagus, the gastric examination and transpyloric passage of the capsule is conducted under magnetic steering, and then examination is continued in the small bowel under intestinal peristalsis.

ELIGIBILITY:
Inclusion Criteria:

* With or without gastrointestinal complaints
* Scheduled to undergo a capsule endoscopy for both stomach and small bowel
* Signed the informed consents before joining this study

Exclusion Criteria:

* Dysphagia or symptoms of gastric outlet obstruction, suspected or known intestinal stenosis, overt gastrointestinal bleeding, history of upper gastrointestinal surgery or abdominal surgery altering gastrointestinal anatomy
* Refused abdominal surgery to take out the capsule in case of capsule retention
* Implanted pacemaker, except the pacemaker is compatible with MRI
* Other implanted electromedical devices or magnetic metal foreign bodies
* Pregnancy or suspected pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China

REFERENCES:
- [Derived] Jiang B, Qian YY, Pan J, Jiang X, Wang YC, Zhu JH, Zou WB, Zhou W, Li ZS, Liao Z. Second-generation magnetically controlled capsule gastroscopy with improved image resolution and frame rate: a randomized controlled clinical trial (with video). Gastrointest Endosc. 2020 Jun;91(6):1379-1387. doi: 10.1016/j.gie.2020.01.027. Epub 2020 Jan 22. PMID 31981648

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.45 (13.51) | 48.58 (14.24) | 48.51 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 24 | 23 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 40 | 80
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 40 | 40 | 80
Indication [Count of Participants; unit: Participants]
  Abdominal pain or distension | 20 | 19 | 39
  Acid reflux or nausea/vomit | 5 | 5 | 10
  Chronic diarrhea | 6 | 4 | 10
  Physical examination | 9 | 12 | 21
Helicobacter pylori (Hp) infection [Count of Participants; unit: Participants] | 7 | 7 | 14
History of abdominal surgery, smoking and drinking [Count of Participants; unit: Participants]
  History of abdominal surgery | 4 | 3 | 7
  Smoking history | 7 | 5 | 12
  Drinking history | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Circumferential Visualization of the Z-line
Description: Circumferential visualization of the Z-line is defined by quadrants as follows: less than 2 quadrants (< 50%) of the Z line observed; at least 2 quadrants (50%-75%) observed; at least 3 quadrants (>75%) observed; and entire Z line (100%) observed.
Time Frame: Through end of examination, up to 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
Number analyzed (Participants) | 40 | 40
Participants
  100% of Z-line | 0 | 5
  ≥50% of Z-line | 5 | 7
  <50% of Z-line | 12 | 12
  0% of Z-line | 23 | 16

2. Secondary Outcome: Detection Rate of Duodenal Papilla
Description: Detection rate of duodenal papilla means the percentage of patients with at least one image of duodenal papilla was obtained
Time Frame: up to 2 days after the examination
Measure: Count of Participants; unit: Participants
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
Number analyzed (Participants) | 40 | 40
Participants | 3 | 6

3. Secondary Outcome: Gastric Examination Time (GET)
Description: Record the time taken for endoscopist to finish the gastric examination for primary anatomical landmarks twice (cardia, fundus, body, angulus, antrum and pylorus).
Time Frame: Through end of examination, up to 30 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
Number analyzed (Participants) | 40 | 40
minutes | 7.78 (0.97) | 5.24 (0.74)

4. Secondary Outcome: Manipulation Performance Score of the MCCG
Description: The performance of maneuverability is assessed using a semi-quantitative score related to the fluency, stability and comfortableness for examination procedure. Fluency is mainly reflected on the response speed to operation and smoothness of video playing. Stability is about the ability of holding the position for a long enough time and the real-time viewing of all images. comfortableness is the operator's sensation about manipulative force and fatigue degree. Maneuverability score was defined as a total scale of 3 to 15 calculated by adding up each evaluation index score above, and each index was graded from 1 to 5, with 1 as the worst and 5 as the best.
Time Frame: up to 10 minutes after the examination
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
Number analyzed (Participants) | 40 | 40
score on a scale
  Fluency | 3.04 (0.51) | 4.59 (0.42)
  Comfortableness | 3.16 (0.45) | 4.51 (0.43)
  Stability | 3.84 (0.55) | 4.17 (0.50)
  Total score | 10.05 (1.04) | 13.28 (0.9)

5. Secondary Outcome: Image Quality Score (Mainly Focus on Clarity)
Description: Assess Image quality grade ranged from 1 to 10 (1, the worst quality; 10, the quality of the best image captured by EGD).
Time Frame: up to 30 minutes after the examination
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
Number analyzed (Participants) | 40 | 40
score on a scale | 7.90 (0.61) | 8.63 (0.57)

6. Secondary Outcome: The Number of Images Captured for Esophagus and Z-line
Description: The number of images captured by MCCG for esophagus and Z-line.
Time Frame: up to 30 minutes after the examination
Measure: Median (Inter-Quartile Range); unit: images
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
Number analyzed (Participants) | 40 | 40
images
  The number of images captured for esophagus | 97 [42 to 160.25] | 171 [81.25 to 409.25]
  The number of images captured for Z-line | 0 [0 to 2.75] | 2 [0 to 13.00]

7. Secondary Outcome: Number of Participants With Lesions in Upper Gastrointestinal Tract
Description: calculate the number of participants with lesions in different part of upper gastrointestinal tract (esophagus, stomach, duodenum, jejunoileum), and preliminarily evaluate the diagnostic efficacy of the new-generation MCCG.
Time Frame: up to 2 days after the examination
Measure: Count of Participants; unit: Participants
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
Number analyzed (Participants) | 40 | 40
Participants
  Inflammation | 25 | 24
  Focal lesions | 12 | 13
  normal | 3 | 3

8. Secondary Outcome: Transit Time of MCCG in the Gastrointestinal Tract and Total Running Time
Description: Assess the transit time of MCCG in the gastrointestinal tract (stomach and small bowel), and record the total running time from starts take images to ends.
Time Frame: up to 2 days after the examination
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
Number analyzed (Participants) | 40 | 40
minutes
  Gastric transit time (min) | 53.09 [22.88 to 90.84] | 48.35 [19.09 to 78.83]
  Small-bowel transit time (min) | 327.60 [260.73 to 394.55] | 297.22 [239.68 to 369.27]
  Total running time (min) | 702.83 [648.47 to 856.10] | 1001.99 [774.42 to 1207.38]

9. Secondary Outcome: Cleansing Level Score of Z-line Area
Description: The bubbles/saliva on the Z line area will be scored as follows: 0 = no bubbles/saliva on the Z line area;1 = a few bubbles/saliva on the Z line area; 2= increased amount of bubbles/saliva on the Z line area; 3 = severe bubbles/saliva on the Z line area.
Time Frame: Through end of examination, up to 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
Number analyzed (Participants) | 40 | 40
Participants
  No bubbles | 13 | 11
  A few bubbles | 18 | 22
  Increased amount of bubbles | 7 | 5
  Severe bubbles | 2 | 2

10. Secondary Outcome: The Incidence of Adverse Events (The Safety of MCCG)
Description: The presence of adverse events within two weeks aftter swallowing MCCG will be recorded.
Time Frame: up to 2 weeks after the examination
Measure: Count of Participants; unit: Participants
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
Number analyzed (Participants) | 40 | 40
Participants | 0 | 0

11. Secondary Outcome: Transit Time of MCCG in Esophagus
Description: Assess the transit time of MCCG in esophagus from starts take images to ends.
Time Frame: up to 2 days after the examination
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
Number analyzed (Participants) | 40 | 40
seconds | 59.5 [24.75 to 82.75] | 44.5 [23.0 to 107.5]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: capsule retention, aspiration of the capsule, severe choking cough and death.
Arm/Group | The First-generation MCCG Group | The Second-generation MCCG Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT03977935/Prot_SAP_000.pdf